CLINICAL TRIAL: NCT04975672
Title: Efficacy of Myofunctional Therapy in Class II Patients With Functional Orthopedic Appliances. ECA
Brief Title: Efficacy of Myofunctional Therapy in Class II Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Sulma Milena Suarez, principal investigator, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2021-03-01; First posted 2021-07-23 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Efficacy; Myofunctional Therapy; Orthopedics
Keywords: Efficacy; Myofunctional Therapy; Dentofacial Orthopedics
MeSH Terms: interventions — Orthopedic Procedures

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two parallel arms
Who Masked: Outcomes Assessor
Masking Description: The operator responsible for making measurements of tongue position, mandibular advancement, orofacial muscle contraction, chin muscle activity, will be blinded to the assignment. A previous training will be carried out with an instruction manual for the clinical evaluation process
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, with myofunctional therapy and SN1 functional orthopedic appliances (Experimental): The participant will receive a session of myofunctional therapy every month, for 9 months. In this group, a series of procedures and techniques are carried out to create and mechanize muscular and orofacial patterns at rest and in function, eliminate habits, correct muscular imbalance, improve the aesthetics of the patient and normalize the functions of the stomatognathic system.
  Interventions: Other: Myofuncional Therapy
- Group 2, without myofunctional therapy and SN1 functional orthopedic appliances. (Experimental): Once the investigation is finished, the patient will decide whether or not to perform myofunctional therapy one every month, for 9 months.
  Interventions: Other: Myofuncional Therapy

INTERVENTIONS:
Other: Myofuncional Therapy — Group 1, with myofunctional therapy and SN1 functional orthopedic appliances The participant underwent a myofunctional therapy session every month, for 9 months. In this group, a series of procedures and techniques are carried out to create and mechanize muscular and orofacial patterns at rest and in function, eliminate habits, correct muscular imbalance, improve the aesthetics of the patient and normalize the functions of the stomatognathic system. The myofunctional therapy performed will be by an expert speech therapist
  Other Names: Orthopedics

SUMMARY:
Randomized clinical trial , with a sample of 60 children with atypical swallowing, class II and with SN1 orthopedic appliances these patients were randomly divided into, group 1: 30 patients with SN1 orthopedic appliances and myofunctional therapy and group 2: 30 patients with SN1 orthopedic appliances and without myofunctional therapy.

DETAILED DESCRIPTION:
Randomized clinical trial with two parallel arms, on a sample of 60 children with atypical swallowing, class II and with SN1 orthopedic appliances, these patients were randomly divided into, group 1: 30 patients with SN1 orthopedic appliances and myofunctional therapy and group 2: 30 patients with SN1 orthopedic appliances and without myofunctional therapy for the study. Both groups carried out the evaluation of the protocol that included: 1) evaluation of the dental occlusion class and skeletal classification 2) swallowing function test using the Payne technique; 3) Mioscaner analysis to measure perioral forces, i.e. tongue extension force, lip pressure, masseter contraction force.

ELIGIBILITY:
Inclusion Criteria:

* the inclusion criteria the participants will be between

  * 8 and 10 years old
  * mixed dentition
  * canine class II diagnosis and 2 to 4 mm
  * molar according to Angle and overjet between 4 to 6 mm

Exclusion Criteria:

* Patients with systemic involvement

  * congenital malformations
  * facial deformities
  * Open bite
  * oral breathing
  * finger sucking habit will be excluded

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-12-22 (Estimated); Primary Completion 2022-12-22 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapy Efficacy / Tongue Position | 9 months
  Lingual projection force
41 / 5000 Resultados de traducción Efficacy of therapy / mandibular advancement | 9 months
  It induces changes in the position of the mandibular bone towards a more advanced position
Muscle contraction | 9 months
  Physiological process in which the muscles develop tension and are shortened or stretched by a stimulus
Contraction of the masseter muscles and muscle activity of the chin | 9 months
  101 / 5000 Resultados de traducción Physiological process in which the muscles develop tension and are shortened or stretched by a stimulus

IPD SHARING:
Plan to Share IPD: No